CLINICAL TRIAL: NCT02586935
Title: A Randomized Placebo-controlled Trial of Tideglusib vs. Placebo in the Treatment of Adolescents With Autism Spectrum Disorders (ASD)
Brief Title: Tideglusib vs. Placebo in the Treatment of Adolescents With Autism Spectrum Disorders
Acronym: TIDE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: McMaster University (Other); Western University, Canada (Other); Unity Health Toronto (Other); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TIDE-06-2015
Record Dates: First submitted 2015-10-16; First posted 2015-10-27 (Estimated); Last update posted 2025-07-16 (Actual); Status verified 2018-05

CONDITIONS: Autism Spectrum Disorders
Keywords: ASD; Autism
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — tideglusib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tideglusib (Active Comparator)
  Interventions: Drug: Tideglusib
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tideglusib — Administered orally after dispersion in approximately 100 ml of water at dose levels of 400 to 1000 mg
  Arms: Tideglusib
Other: Placebo — Administered orally after dispersion in approximately 100 ml of water
  Arms: Placebo

SUMMARY:
This study will examine the safety and efficacy of tideglusib vs. placebo for the treatment of core symptom domains in adolescents with Autism Spectrum Disorders

DETAILED DESCRIPTION:
There are no pharmacologic treatments available for social function deficits in individuals with Autism Spectrum Disorders (ASD). The data for pharmacologic treatment of repetitive behaviours in this disorder has also become difficult to interpret given that the last two large multisite trials of selective serotonin re-uptake inhibitors (SSRIs) in autism are reported to be negative for the treatment of repetitive behaviours. Only the associated symptom of irritability has 2 drugs with Food and Drug Administration (FDA) indications, whereas no systematic data exists on the pharmacologic treatment of anxiety in ASD, and response rates to stimulants for hyperactivity are lower than what is seen in Attention Deficit Hyperactivity Disorder (ADHD). In addition, there are no biological markers of treatment response identified in this population at this point. This study will examine the potential efficacy and safety of tideglusib for core and associated symptom domains of autism, and will explore biological markers of safety and treatment response. As there is no juvenile toxicity published in the animal model, we will limit the age range to 12 years of age and older.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients 12-17 years of age inclusive with a mental age equivalent ≥ 18 months at Screening.
2. Weigh a minimum of 30 kg (the 3rd percentile for 12 years of age)
3. Meet Diagnostic and Statistical Manual of Mental Disorders. Diagnostic and Statistical Manual (DSM-5) criteria will be established by a clinician with expertise with individuals with ASD.
4. Have a Clinician's Global Impression-Severity (CGI-S) score ≥ 4 (moderately ill) at Screening.
5. If already receiving stable concomitant medications affecting behaviour, have stable regimens with no changes during the preceding 1 month prior to Screening (with the exception of fluoxetine, where a period of 6 weeks is needed), and will not electively initiate new or modify ongoing medications for the duration of the study
6. If already receiving stable non-pharmacological educational and behavioural interventions, have continuous participation during the preceding 3 months prior to Screening, and not electively initiate new or modify ongoing interventions for the duration of the study
7. Have normal physical examination and laboratory test results at Screening. If abnormal, the finding(s) must be deemed clinically insignificant by the Investigator.
8. Ability to obtain written informed consent from the participant, if developmentally appropriate. If a participant does not have the capacity to consent, ability to obtain assent (if developmentally appropriate), as well as written informed consent from their parent(s)/legal guardian.

Exclusion Criteria:

1. Patients with a primary psychiatric diagnosis other than ASD
2. Pregnant female patients; sexually active female patients on inadequate birth control.
3. Patients with known phosphatase and tensin homolog (PTEN) mutations as they are unlikely to respond to this medication
4. Patients with a serious medical condition that, based on Investigator judgment, might interfere with the conduct of the study, confound interpretation of the study results, or endanger their own well-being. Patients with evidence of any significant hematological, endocrine, cardiovascular (including uncorrected symptomatic congenital heart disease), respiratory, renal, hepatic, or gastrointestinal disease, not including mild common pediatric diseases in these areas that are stable (e.g. mild asthma, constipation, etc.).
5. Patients with unstable epilepsy (i.e. seizures occurring within the last 6 months), or patients with epilepsy who are not on stable doses of antiepileptic medications (i.e. dose changes within the last 3 months).
6. Patients with hypersensitivity to tideglusib or any components of its formulation.
7. Patients unable to tolerate venipuncture procedures for blood sampling.
8. Patients actively enrolled in another intervention study.
9. Patients who have elevated liver enzymes ≥ 3 times the normal amount before the study begins.
10. Patients who have serum creatinine of >150 μmol/L and creatinine clearance ≤60ml/m (according to Cockcroft-Gault formula) at Screening.
11. Patients taking strong CYP3A4 inhibitors (e.g. clarithromycin, telithromycin, ketoconazole, itraconazole, posaconazole, nefazodone, indinavir, ritonavir)
12. Inability to speak and understand English sufficiently enough to allow for the completion of all study assessments (parent; patient, if verbal).

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2016-02-10 (Actual); Primary Completion 2018-02-25 (Actual); Study Completion 2018-02-25 (Actual)

PRIMARY OUTCOMES:
Effect of tideglusib vs. placebo on measures of social engagement/withdrawal | 12 weeks
  This will be measured by the Aberrant Behavior Checklist (ABC) - Lethargy / Social Withdrawal Subscale

SECONDARY OUTCOMES:
Efficacy of tideglusib vs. placebo on measures of repetitive behaviours | 12 weeks
  This will be measured by the Child Yale-Brown Obsessive Compulsive Scale (CY-BOCS)
Efficacy of tideglusib vs. placebo on measures of repetitive behaviours | 12 weeks
  This will be measured by the Repetitive Behavior Scale (RBS-R)
Efficacy of tideglusib vs. placebo on measures of social function | 12 weeks
  This will be measured by the Vineland Adaptive Behavior Scales, Second Edition (VABS-II) - Socialization Domain
Safety and tolerability of tideglusib in adolescents with ASD | 12 weeks
  This will be measured by the Clinical Global Impressions - Improvement Scale - Global (CGI-I-Global)
Safety and tolerability of tideglusib in adolescents with ASD | 12 weeks
  This will be measured by the Safety Monitoring Uniform Report Form (SMURF)
Pharmacokinetic (PK) parameters in this age group | 12 weeks
  This will be completed by measuring / calculating Cmax (Peak Plasma Concentration)
Pharmacokinetic (PK) parameters in this age group | 12 weeks
  This will be completed by measuring / calculating C0-6 (Steady State Plasma Concentration)
Pharmacokinetic (PK) parameters in this age group | 12 weeks
  This will be completed by measuring / calculating Area Under the Curve (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Evdokia Anagnostou, M.D., Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital; Terry Bennett, M.D., Principal Investigator — MacMaster University, Offord Centre for Child Studies; Robert Nicolson, M.D., Principal Investigator — University of Western Ontario, Lawson Health Research Institute
Locations (3):
- Canada (3):
  - McMaster University, Offord Centre for Child Studies, Hamilton, Ontario
  - University of Western Ontario, Lawson Health Research Institute, London, Ontario
  - Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No